CLINICAL TRIAL: NCT07075536
Title: A Web-based Contraceptive Decision Support Tool for Individuals With Health Conditions: A Cluster Randomized Controlled Trial With Mixed Methods
Brief Title: A Web-Based Tool to Help People With Health Conditions Make Contraceptive Decisions
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); DARTNet Institute (Other Government)
Responsible Party: Principal Investigator, Justine Wu, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00234187; 5R01HD110570-02 (NIH)
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Contraceptive Usage; Contraceptive Behavior; Chronic Disease; Chronic Condition; Chronic Conditions, Multiple
Keywords: Contraceptive Use; Contraceptive decision making; Shared Decision Making; Person-Centered Contraceptive Counseling; Decisional Conflict; Web-Based Tool
MeSH Terms: conditions — Contraception Behavior; Chronic Disease; Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel cluster randomized controlled trial using mixed methods (the collection and integration of quantitative and qualitative data) to compare the intervention (My Health My Choice decision tool) to usual contraceptive care in 14 outpatient clinics that provide contraceptive services. Randomization occurs at the clinic level to prevent contamination across patients and clinicians in the same clinic.
Who Masked: Outcomes Assessor
Masking Description: The lead biostatistician will generate the allocation sequence and assign clinics to the intervention arm or usual care arm. To prevent unequal distribution of clinics that have greater expertise in contraceptive care, clinics with family planning specialists will be balanced between the two arms. Because of the cluster RCT design, allocation concealment is impractical. To minimize the risk of recruitment bias, differential dropouts, and bias, group assignments will be revealed to patient and clinician participants only after they have been consented and taken the baseline survey. The study team and statistical team will be blinded to group assignment when evaluating outcomes. This approach is consistent with the Ottawa Statement on the Ethical Design and Conduct of Cluster Randomized Trials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- My Health, My Choice Contraceptive Decision Tool (Experimental): Participants in the intervention arm will use a web-based, password-protected contraceptive decision support tool (My Health My Choice) prior to a clinic visit with a licensed clinician who provides contraceptive care (CNM, DO, MD, NP, PA).
  Interventions: Behavioral: My Health, My Choice Web-Based Contraceptive Decision Tool
- Usual Contraceptive Care (Placebo Comparator): Participants will receive usual contraceptive care from a licensed provider (CNM, DO, MD, NP, PA).
  Interventions: Behavioral: Usual Contraceptive Care

INTERVENTIONS:
Behavioral: My Health, My Choice Web-Based Contraceptive Decision Tool — The My Health My Choice decision tool is a web-based interactive tool designed to educate patients with health conditions about their contraceptive options, elicit their personal preferences and contraceptive concerns, and help them prepare for a contraceptive discussion with their clinician. Patients can compare features of different contraceptive methods side-by-side and grouped by medical risk according to the Center for Disease Control and Prevention U.S. Medical Eligibility Criteria (US MEC). The tool generates an individualized Birth Control Summary for each patient user that records their "contraceptive favorites" and their questions for the clinician. Clinicians can use the Clinician Version of the tool to review the patient's Birth Control Summary and their medical eligibility for different contraceptive methods per the US MEC guidelines.
  Arms: My Health, My Choice Contraceptive Decision Tool
Behavioral: Usual Contraceptive Care — Participants will attend clinic visits per routine. Clinicians proceed with usual contraceptive care. All study activities and incentives for participants in the usual contraceptive care arm are the same as for participants in the intervention arm except for those related to the intervention itself.
  Arms: Usual Contraceptive Care

SUMMARY:
Among people who do not want to get pregnant, some do not use any birth control. This is also called contraceptive nonuse. Common reasons for contraceptive nonuse include concerns about birth control safety or side effects. People with health conditions, such as diabetes or high blood pressure, also report worries about how different birth control methods might affect their health condition or medicines.

The goal of this clinical trial is to learn if a web tool called My Health, My Choice helps people with health conditions understand their birth control options and choose birth control that is right for them. The study will also look at the medical safety of birth control methods that participants decide to use. The main questions it aims to answer are:

• Does the My Health My Choice tool lower the number of participants who do not use any birth control method? (contraceptive nonuse)

In other words, does the My Health My Choice tool increase the number of participants who use any birth control method? (contraceptive use)

Participants who use the My Health, My Choice tool before a clinic visit with their clinician (Intervention Group) will be compared to participants who only go to a clinic visit with their clinician (Usual Care Group).

For this study, a "clinician" is any licensed health care provider who counsels about birth control, prescribes birth control, and/or inserts birth control devices.

All participants will:

* Complete 4-5 online surveys that take 5-10 minutes each, over a 3 month time period
* Be asked to go to a scheduled clinic visit with their health care provider
* A small group of participants (about 30) will be invited to a 1 hour exit interview

Participants in the intervention arm will be asked to:

• Use the My Health My Choice tool before their clinic visit

DETAILED DESCRIPTION:
Fourteen outpatient clinics in the United States that provide birth control services, including primary care and obstetrics and gynecology clinics, will be enrolled. Each clinic will be randomly assigned to the My Health My Choice Group (intervention group) or the Usual Care group. Only patients who receive health care at enrolled clinics are eligible for study participation.

Participants must be aged 18-49 years, read English, fertile (able to get pregnant), have at least one index health condition, characteristic or medication usage (full list of 60+ eligible conditions, characteristics, and 50+ medications available upon request); and want to talk about birth control at an upcoming clinic visit with their clinician.

Eligible participants will be enrolled over the phone. Enrolled participants will complete a baseline electronic survey about their demographics, health history, contraceptive use, and contraceptive knowledge before learning which study group they are in.

Study Activities for Participants in the Intervention Arm Only:

* Before their scheduled clinic visit, open and use the My Health My Choice tool via a password-protected weblink on a mobile device, computer
* Complete a brief electronic survey about their experience using the My Health My Choice web tool.

Study Activities for All Participants:

* Go to their scheduled clinic visit with their clinician
* Complete a survey shortly after the clinic visit
* Complete a survey 1 month after the clinic visit
* Complete a survey 3 months after the clinic visit

All surveys take about 5-10 minutes to complete. About 30 participants across all clinic sites will be asked to do an optional 1 hour exit interview by phone or teleconference.

Clinicians who provide contraceptive care, including residents who have finished their intern year, are eligible to participate. Eligible clinicians include doctors, nurse practitioners, physician assistants, and certified nurse midwives. Enrolled clinicians will complete a brief baseline and exit survey about their contraceptive counseling, the type of contraceptive methods they provide, and their contraceptive knowledge.

Activities for All Clinicians

* Complete a baseline survey
* Complete an exit survey
* Provide care to enrolled patients at their scheduled visits
* Complete a brief survey after each visit with an enrolled patient

Activities for Clinicians in the Intervention Arm Only

• Before or during the scheduled clinic visit, open and use Clinician Version of the My Health My Choice tool via a password-protected weblink on a mobile device, computer

The Clinician Version of the My Health My Choice has information to help clinicians counsel patients with health conditions about the safety of different birth control methods. Clinicians can also review the "Birth Control Summary" of enrolled patients before or during the clinic visit.

All clinician surveys take 3-10 minutes to complete. About 30 clinician participants across all clinic sites will be asked to participate in an optional 1 hour exit interview by phone or teleconference.

After patients exit the study, an electronic health record (EHR) review will be done to find out if participants got birth control prescriptions or birth control devices during the study. The EHR review also includes checking if participants report plans to get permanent birth control (tubal sterilization for themselves or vasectomy for their partners).

The primary and secondary outcomes are patient-reported or patient-related outcomes. There are no primary or secondary outcomes for clinicians.

The study aims to enroll 725 patients and 70 clinicians (795 in total).

ELIGIBILITY:
Patient Inclusion Criteria:

* Between the ages of 18 and 49
* Assigned female sex at birth, regardless of gender identity
* Presumed to be fertile (have an intact uterus/tube/ovary; premenopausal)
* Have at least one index health condition, characteristic or medication usage (full list of 60+ eligible conditions, characteristics, and 50+ medications available upon request); and want to talk about birth control at an upcoming clinic visit with their clinician
* Able to read in English
* Access to mobile phone, computer, or tablet with internet capabilities
* Not currently pregnant
* Desire to talk to their clinician about starting, switching, or adding a contraceptive method for the purpose of preventing pregnancy

Patient Exclusion Criteria:

* Trying to get pregnant in the next 12 months
* Presumed infertile for any surgical or medical reason (e.g., postmenopausal, hysterectomy, chemotherapy)

There are additional clarifications regarding patient eligibility, such as a full list of eligible medical diagnoses and medicines, that can be found in the protocol.

Clinician Inclusion Criteria:

• Any licensed clinician who provides contraceptive care at a participating clinic, including physicians, physician assistants, certified nurse midwives, nurse practitioners. (For clinicians, there are no restrictions based upon age, gender identify or sex).

Clinician Exclusion Criteria:

• Physician interns (PGY-1) are not eligible

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 795 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who report contraceptive nonuse at 3 months | Baseline, 1 month, and 3 months after the clinic visit
  This is a binary outcome (yes/no) that will be assessed at baseline, 1 month, and 3 months after the clinic visit. Participants will report use or nonuse of a contraceptive method in the last month. Contraceptive methods include all non-prescription methods, prescription methods, intrauterine devices (IUDs), the implant, tubal ligation/surgery, and vasectomy of their partner.
  If patients report use of the cervical cap, condoms, diaphragm, spermicides, vaginal gel, or withdrawal, their outcome will be determined by whether they used the method at last intercourse in the prior month.
  Only patients who did not want to get pregnant in the last month will be included in the calculation of this outcome.

SECONDARY OUTCOMES:
Medical Eligibility Risk (MER) Category among participants who report contraceptive method use | Baseline, 1 month, and 3 months
  The Medical Eligibility Risk (MER) Category will be determined for participants who report contraceptive use at baseline, 1 month, and 3 months. Based upon the patient's health history and reported contraceptive method, two contraceptive experts blinded to patient assignment will assign the MER per the U.S. Medical Eligibility Criteria Guidelines. This is a categorical measure with four MER Categories:
  * Category 1: the method can be used without restriction because there are no theoretical or proven risks
  * Category 2: the method can be used because the advantages outweigh any theoretical or proven risks
  * Category 3: in general, the method should be avoided because the theoretical or proven risks of a contraceptive method usually outweigh any advantages of use.
  * Category 4: the method should not be used because the theoretical or proven risks outweigh any advantages.

CONTACTS AND LOCATIONS:
Overall Officials: Justine P Wu, MD, MPH, Principal Investigator — Department of Family Medicine, University of Michigan
Locations (18):
- United States (18):
  - University of Arizona College of Medicine - Phoenix Department of Family, Community and Preventive Medicine - Research Division & Arizona Developing Experience with Practice-Based Research Network (PBRN) Studies, Phoenix, Arizona
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Full Circle Health Family Medicine Residency of Idaho - Nampa Program, Nampa, Idaho
  - University of Kansas Medical Center Department of Family Medicine & Community Health, Kansas City, Kansas
  - MaineHealth Primary Care - Family Medicine - Sanford, Sanford, Maine
  - Boston Medical Center's Department of Family Medicine, Boston, Massachusetts
  - Department of Family Medicine Research Office, Ann Arbor, Michigan
  - Von Voigtlander Women's Hospital Obstetrics and Gynecology clinic, Ann Arbor, Michigan
  - Michigan State University Health Care Family Medicine, East Lansing, Michigan
  - WMed Health Family Medicine - Crosstown Parkway, Kalamazoo, Michigan
  - Munson Family Practice Center, Traverse City, Michigan
  - Ypsilanti Health Clinic, Ypsilanti, Michigan
  - Rutgers Robert Wood Johnson Medical School - Family Medicine at Monument Square, New Brunswick, New Jersey
  - Capital Health Family Medicine, Pennington, New Jersey
  - Mountain Area Health Education Center (MAHEC) Family Health Center at Biltmore, Asheville, North Carolina
  - Cleveland Clinic - Complex Family Planning Clinics: Main Campus, Beachwood Family Health Center, Westlake Medical Campus, Cleveland, Ohio
  - Ascent Center for Reproductive Health at the University of Utah, Salt Lake City, Utah
  - West Virginia University School of Medicine - Department of Family Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
All quantitative IPD collected during the trial will be de-identified and made available per the time frame and access criteria described below. The full study protocol and statistical analysis plan will also be published in an open-access peer reviewed journal and made available upon request at FAMMED-BirthControlStudy@med.umich.edu.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All de-identified quantitative IPD and supporting information will be available beginning 1 year after publication of trial findings and for an additional 36 months. After this 36 month time period, the quantitative data will be available in the University of Michigan's Deep Blue Data Repository indefinitely, but without investigator support other than deposited metadata.
Access Criteria: All de-identified quantitative IPD and supporting information will be made available without cost to researchers and analysts upon request to FAMMED-BirthControlStudy@med.umich.edu. These requests will be honored only under a data sharing agreement that requires the user's commitment to: 1) use the data only for research purposes; 2) not identify any individual participant; 3) secure the data using appropriate computer technology; and 4) destroy or return the data after analyses are completed. The information provided to users will not be used for commercial purposes and will not be redistributed to third parties. In addition to dissemination of findings via communication channels such as speaking engagements and publications, these data also may be distributed via online databases, spreadsheets, and other electronic media.

REFERENCES:
- [Background] Campbell MK, Elbourne DR, Altman DG; CONSORT group. CONSORT statement: extension to cluster randomised trials. BMJ. 2004 Mar 20;328(7441):702-8. doi: 10.1136/bmj.328.7441.702. No abstract available. PMID 15031246
- [Background] Dehlendorf C, Henderson JT, Vittinghoff E, Grumbach K, Levy K, Schmittdiel J, Lee J, Schillinger D, Steinauer J. Association of the quality of interpersonal care during family planning counseling with contraceptive use. Am J Obstet Gynecol. 2016 Jul;215(1):78.e1-9. doi: 10.1016/j.ajog.2016.01.173. Epub 2016 Jan 28. PMID 26827879
- [Background] Thompson R, Manski R, Donnelly KZ, Stevens G, Agusti D, Banach M, Boardman MB, Brady P, Colon Bradt C, Foster T, Johnson DJ, Li Z, Norsigian J, Nothnagle M, Olson AL, Shepherd HL, Stern LF, Tosteson TD, Trevena L, Upadhya KK, Elwyn G. Right For Me: protocol for a cluster randomised trial of two interventions for facilitating shared decision-making about contraceptive methods. BMJ Open. 2017 Oct 22;7(10):e017830. doi: 10.1136/bmjopen-2017-017830. PMID 29061624
- [Background] Murray DM, Blistein JL. Methods to reduce the impact of intraclass correlation in group-randomized trials. Eval Rev. 2003 Feb;27(1):79-103. doi: 10.1177/0193841X02239019. PMID 12568061
- [Background] Murphy DM. Planning the Trial. Design and Analysis of Group-Randomized Trials. Oxford University Press; 1998:19-65
- [Background] Weijer C, Grimshaw JM, Eccles MP, McRae AD, White A, Brehaut JC, Taljaard M; Ottawa Ethics of Cluster Randomized Trials Consensus Group. The Ottawa Statement on the Ethical Design and Conduct of Cluster Randomized Trials. PLoS Med. 2012;9(11):e1001346. doi: 10.1371/journal.pmed.1001346. Epub 2012 Nov 20. PMID 23185138
- [Background] Stacey D, Legare F, Boland L, Lewis KB, Loiselle MC, Hoefel L, Garvelink M, O'Connor A. 20th Anniversary Ottawa Decision Support Framework: Part 3 Overview of Systematic Reviews and Updated Framework. Med Decis Making. 2020 Apr;40(3):379-398. doi: 10.1177/0272989X20911870. PMID 32428429
- [Background] Kang MM, Guetterman TC, Prussack JK, Ursu A, Wu JP. Contraceptive Care for Women With Medical Conditions: A Qualitative Study to Identify Potential Best Practices for Primary Care Physicians. Fam Med. 2019 Jul;51(7):559-566. doi: 10.22454/FamMed.2019.499467. PMID 31287901
- [Background] Dehlendorf C, Fitzpatrick J, Fox E, Holt K, Vittinghoff E, Reed R, Campora MP, Sokoloff A, Kuppermann M. Cluster randomized trial of a patient-centered contraceptive decision support tool, My Birth Control. Am J Obstet Gynecol. 2019 Jun;220(6):565.e1-565.e12. doi: 10.1016/j.ajog.2019.02.015. Epub 2019 Feb 11. PMID 30763545
- [Background] Chor J, Rankin K, Harwood B, Handler A. Unintended pregnancy and postpartum contraceptive use in women with and without chronic medical disease who experienced a live birth. Contraception. 2011 Jul;84(1):57-63. doi: 10.1016/j.contraception.2010.11.018. Epub 2011 Jan 20. PMID 21664511
- [Background] Judge CP, Zhao X, Sileanu FE, Mor MK, Borrero S. Medical contraindications to estrogen and contraceptive use among women veterans. Am J Obstet Gynecol. 2018 Feb;218(2):234.e1-234.e9. doi: 10.1016/j.ajog.2017.10.020. Epub 2017 Oct 27. PMID 29111146
- [Background] ACOG Practice Bulletin No. 206 Summary: Use of Hormonal Contraception in Women With Coexisting Medical Conditions. Obstet Gynecol. 2019 Feb;133(2):396-399. doi: 10.1097/AOG.0000000000003073. PMID 30681537
- [Background] Fox E, Reyna A, Malcolm NM, Rosmarin RB, Zapata LB, Frederiksen BN, Moskosky SB, Dehlendorf C. Client Preferences for Contraceptive Counseling: A Systematic Review. Am J Prev Med. 2018 Nov;55(5):691-702. doi: 10.1016/j.amepre.2018.06.006. PMID 30342632
- [Background] Russo JA, Chen BA, Creinin MD. Primary care physician familiarity with U.S. medical eligibility for contraceptive use. Fam Med. 2015 Jan;47(1):15-21. PMID 25646873
- [Background] Wu JP, Gundersen DA, Pickle S. Are the Contraceptive Recommendations of Family Medicine Educators Evidence-Based? A CERA Survey. Fam Med. 2016 May;48(5):345-52. PMID 27159092
- [Derived] Palazzolo B, Aikens JE, Sen A, Guetterman TC, Buis LR, Dalton VK, Zikmund-Fisher BJ, Mabachi N, Kang M, Dehlendorf C, Van Sparrentak M, Lutgen CB, Wynn C, Wu JP. A Web-Based Contraception Decision Tool for Individuals With Health Conditions in US Outpatient Clinics: Protocol for a Mixed Methods Cluster Randomized Controlled Trial. JMIR Res Protoc. 2025 Dec 29;14:e71101. doi: 10.2196/71101. PMID 41461082
- See also: My Health My Choice Study Website — https://sites.google.com/umich.edu/my-health-my-choice-study/home?authuser=1